CLINICAL TRIAL: NCT06949813
Title: Preventing Maternal Mood, Anxiety, and Trauma Symptoms After Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-2499; 1R34MH133685-01A1 (NIH)
Record Dates: First submitted 2024-11-01; First posted 2025-04-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Anxiety in Pregnancy; Mood Disorder Due to Specified Medical Condition
Keywords: perinatal mood and anxiety disorders; cesarean delivery; Single session immersive intervention; Randomized Controlled Trial
MeSH Terms: conditions — Anxiety Disorders | interventions — Cesarean Section

STUDY DESIGN:
Intervention Model Description: 2:1:1 randomization allocation of 3 study groups. Intervention: (N= 40) Participants will be scheduled to receive the 1-hour, single-session CARE intervention administered by a medical and mental health provider trained in the intervention. CARE will consist of psychoeducation and brief immersive exposure to the operating room.
  Interaction Control: (N = 20) Participants will receive a 1-hour, single-session meeting with a nurse educator that will occur within a single patient room on L&D. This condition will provide the same front-line clinician facetime as the treatment condition but will not include the clinical content of the intervention (psychoeducation + exposure).
  Care as Usual Control: (N = 20) Participants will receive all the standard education. The participants will not receive any additional face-to-face interaction with front-line clinicians as part of the study.
Who Masked: Participant
Masking Description: After providing informed consent, participants will be randomized (2:1:1) to condition using an Excel spreadsheet uploaded into a REDCap® database. This will ensure allocation concealment. At the time of consent, patients will be informed that the study involves randomization to one of three conditions, two of which involve a one-hour session with one or more clinicians to prepare the participants for delivery. Participants assigned to BE-OR versus Interaction Control conditions will be informed that they are assigned to a condition in which they receive an intervention but will be masked to whether they were assigned to BE-OR or Interaction Control "intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Intervention: (N= 40) Participants will be scheduled to receive the 1-hour, single-session CARE intervention administered by a medical and mental health provider trained in the intervention. CARE will consist of psychoeducation and brief immersive exposure to the operating room.
  Interventions: Behavioral: BE-OR: Brief Intervention to the Operating Room
- Interaction Control (Experimental): Interaction Control: (N = 20) Participants will receive a 1-hour, single-session meeting with a nurse educator that will occur within a single patient room on L&D. This condition will provide the same front-line clinician facetime as the treatment condition but will not include the clinical content of the intervention (psychoeducation + exposure).
  Interventions: Other: Interaction: Facetime with Clinical Provider
- Care as Usual (No Intervention): Care as Usual Control: (N = 20) Participants will receive all the standard prenatal and CD education. The participants will not receive any additional face-to-face interaction with front-line clinicians as part of the study.

INTERVENTIONS:
Behavioral: BE-OR: Brief Intervention to the Operating Room — See intervention group section for details
  Other Names: CARE-CD: Comfort, Agency, Readiness, Empowerment for Cesarean Delivery
  Arms: Intervention
Other: Interaction: Facetime with Clinical Provider — See Interaction group section for details
  Arms: Interaction Control

SUMMARY:
Perinatal mental health disorders are the most prevalent perinatal comorbidity and are associated with the primary cause of maternal mortality in the United States (US) - suicide. Diagnosis of a high-risk pregnancy and cesarean delivery (CD) are both associated with increased risk for perinatal mood, anxiety, and trauma symptoms (PMATS). There is a deficit in resources and access to mental health treatment for pregnant patients, with some treatments being cost-prohibitive and requiring multiple sessions. Additionally, current approaches to addressing PMATS are reactive rather than preventive. There is evidence in the non-obstetric population that single-session cognitive behavioral therapy interventions targeting anxiety sensitivity (fear of fear) can prevent the development of anxiety and trauma symptoms when individuals are exposed to trauma. The investigators developed a low-cost, 1-hour, single-session prevention intervention that included psychoeducation about anxiety sensitivity, coupled with a brief exposure to the operating room environment and CD procedures. To revise the implementation plan and intervention (CARE: Communication, Agency, Readiness, Empowerment for cesarean delivery [CD]) for use in large L&D units with a broader population of patients, a fully powered multisite randomized control trial (RCT) is needed. Before initiating such a trial, work needs to be done to modify the intervention and implementation through a process of iterative refinement to enhance the acceptability, appropriateness, and feasibility of implementation in L&D units across the country, as well as its efficacy at engaging with the target mechanism (anxiety sensitivity). Using a logic model to guide the iterative refinement process through fast feedback loops and an atmosphere of co-creation, study investigators will gather critical input from stakeholders (individuals with lived experiences, community partners, front-line clinicians, and hospital staff) via 12 workgroups, 12 user-testing design sessions, and repeated engagement with a steering council. Following this refinement process, a treatment development pilot RCT at a large L&D unit will assess the efficacy of CARE for CD by probing engagement with the target mechanism, as well as assess the feasibility of implementation. Finally, the updated logic model and pilot trial results will inform the development of a protocol for a multisite RCT through engagement with expert consultants in a community engagement studio and further feedback from the steering council.

DETAILED DESCRIPTION:
Postpartum mental health disorders disproportionately occur among the 1 million patients with cesarean deliveries (CD) in the United States (US) each year, with 1 in 3 reporting elevated symptoms of postpartum mood, anxiety, and trauma symptoms (PMATS). Brief, single-session interventions that target anxiety sensitivity (AS) through psychoeducation + exposure have been shown to prevent the development of anxiety and trauma symptoms in non-perinatal populations. Thus, a single session AS-targeted intervention involving psychoeducation about AS + in-vivo exposure to the operating room (OR) and CD procedures may be an effective intervention to prevent the development of PMATS. The primary objective of this proposal is to refine and pilot a 1-hour, single-session brief exposure intervention in the OR (CARE) to reduce AS and thus prevent the development of PMATS among a population of patients with high-risk pregnancies and anticipated CD.

The investigators initially developed CARE for implementation in a maternal-fetal care unit at a children's hospital that has 12 beds, an average daily census of 6 patients, and 130 CDs/year. In this unit, the investigators conducted a pilot RCT study of CARE among a population of pregnant patients at very high risk for PMATS (those with anomalous fetuses). Those who received CARE reported 42% less preoperative anxiety and 40% less postpartum anxiety symptoms at 6-8 weeks following delivery, and significantly less opioid use at postoperative days 2-4 than those who received care as usual. While these results demonstrate the promise of the intervention, its scalability to large L&D units and a broader population of patients is not established, and a fully powered, multisite randomized controlled trial (m-RCT) is needed. Before the m-RCT, the intervention must be refined to improve its acceptability, appropriateness, and feasibility for implementation in broader contexts with the desired impact on the target mechanism and outcomes. The proposed project engages in Stage 1A/B activities across three phases. Phase 1 involves a process of iterative refinement using key stakeholder workgroups, user-testing design, and repeated engagement with a steering council (SC) in fast feedback loops to facilitate information flow and foster co-creation. Phase 2 involves the design and implementation of a treatment development trial with an emphasis on feasibility, fidelity, and safety, as well as probing efficacy of engagement with the hypothesized mechanism of CARE (AS) at a single large L&D unit with 50 beds, an average daily census of 34 patients, and 1,000 CDs/year. Phase 3 will involve one additional cycle of rapid iterative refinement to prepare for a future m-RCT with L&D units across the US. Identified future m-RCT site-based investigators and associated administrators will participate in a community engagement studio to refine/co-create a finalized implementation protocol for the m-RCT to take to the SC for final approval.

Specific Aim 1: To enhance the efficacy, responsiveness to diverse populations, scalability, and sustainability of CARE for implementation in large L&D units by engaging in an iterative refinement process guided by an Implementation Research Logic Model (IRLM) framework,12 which allows the team to rapidly iterate based on feedback in Plan-Do-Check-Act cycles using 12 workgroups, 12 user-testing design sessions, and repeated engagement with a SC comprised of stakeholders from across the country (clinicians/hospital staff and those with lived experiences/community partners).

Hypothesis 1: Some barriers and determinants must be addressed to refine CARE and its implementation so that it is acceptable and engages the target mechanism in a diverse population of patients and may be incorporated into workflows on L&D units.

Specific Aim 2: To probe the efficacy of CARE at reducing AS and preventing PMATS using a treatment development trial with high-risk antepartum patients anticipating CD by comparing outcomes among participants randomized to CARE (N=40), Interaction Control (N=20), or Care as Usual Control (N=20) and to establish feasibility, safety, and acceptability of CARE implementation.

Hypothesis 2a: In comparison to patients who receive either control condition, those who receive CARE will have decreased AS before CD.

Hypothesis 2b: Decreased AS before CD will be associated with fewer symptoms of PMATS at 12 weeks postpartum.

Hypothesis 2c: CARE will be administered with high fidelity, yield minimal safety events, and have high acceptability.

Impact Statement: This study is a critical step in preventing PMATS which are among the leading causes of maternal mortality in the US. This study will be the first in a long line of research broadening to additional risk groups, perinatal care settings, and intervention modalities (e.g., virtual reality, nurse- or peer-facilitated).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Patients at 22-37 weeks gestation
* Single or multiple gestation
* Nulliparous or multiparous (with prior vaginal or cesarean delivery)
* Antepartum admission for at least 3 days
* High-risk pregnancy due to maternal/fetal comorbidities
* Anticipated cesarean delivery at the University of Colorado

Exclusion Criteria:

* Lack of capacity to consent
* Medical factors prohibiting participation in the intervention as determined by the inpatient obstetric medical team.
* Anticipated cesarean within 7 days of enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be able to become pregnant, biological female. No exclusion will be made for how a person identifies regarding gender.
Enrollment: 80 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety-sensitivity Index 3 | Baseline
  18-item scale that yields a primary outcome score and subscale scores. Higher scores indicate higher anxiety sensitivity. Minimum score 0. Maximum score 72.
Anxiety-sensitivity Index 3 | Approximately 3 days (range=1-5) after intervention (CARE and interaction control conditions) or approximately 5 days (range = 3-7) after enrollment (care as usual condition)
  18-item scale that yields a primary outcome score and subscale scores. Higher scores indicate higher anxiety sensitivity. Minimum score 0. Maximum score 72.

SECONDARY OUTCOMES:
Adverse Childhood Experience Questionnaire | Baseline
  10-question scale regarding adverse social experiences in childhood. Higher score reflects higher adverse experiences. Minimum score 0. Maximum score 10.
Wijma Delivery Expectancy/Experience Questionnaire | Baseline
  33-item measure of fear of childbirth expectancy. Higher scores are related to higher fear regarding childbirth. Higher scores indicate more fear. Minimum score 0. Maximum score 165.
State-Trait Anxiety Inventory | Baseline
  20-item scale to assess state anxiety symptom intensity. Higher scores indicate more intense anxiety symptoms. Minimum score 20. Maximum score 80.
Columbia Suicide Severity Rating Scale | Baseline
  6-item scale to assess presence of suicidal ideation, plan and intent. Answers are yes or no. With any yes answer indicating some form of suicidality.
Edinburgh postpartum depression scale | Baseline
  10-item scale to assess the presence of depression symptoms in the perinatal period. Higher scores indicate higher incidence of depressive symptoms. Minimum score 0. Maximum score 30.
DSM-5 Cross Cutting Assessment | Baseline
  23-question screening tool developed by the American Psychiatric Association to help clinicians identify symptoms across multiple psychiatric domains. Higher score indicates more adverse symptoms. Minimum score 0. Maximum score 92.
WHO Disability Assessment Schedule (WHODAS 2.0) | Baseline
  World Health Organization Disability Assessment Schedule 2.0 is a 36-question standardized tool to measure health and disability across cultures and diseases, including physical, mental, and substance use disorders. Scale of 1-5 for each question. Minumum score 36. Maximum score 180. The higher the score, higher the disability.
Patient Health Questionnaire-9 | Baseline
  PHQ-9: A nine-question screening tool designed to assess the presence and severity of depression. Score is 0-3 per question. Minimum score 0. Maximum score 27. A score of 10 or more is often used as a clinical cutoff for identifying possible major depression.
Cesarean Section Anxiety Sensitivity (C-SAS) | Baseline
  19-question assessment of anxiety specifically related to events surrounding a cesarean delivery. Score is 1-5 for each question. Minimum score 19. Maximum score 95.
General Anxiety Disorder-7 (GAD-7) | Baseline
  The 7-question screening tool used to assess the severity of generalized anxiety disorder (GAD). 0-3 score per question. Minimum score 0. Maximum score 21. A score of 10 or above is commonly used as a cutoff for identifying potential GAD.
RCADS-25 | Baseline
  25-question questionnaire designed to assess symptoms of anxiety and depression in children and adolescents. Score range 0-3 per question. Minimum score 0. Maximum score 75. The higher the score, the greater the likelihood of clinically significant anxiety or depression.
Cesarean Section Anxiety Sensitivity (C-SAS) | Approximately 3 days (range=1-5) after intervention (CARE and interaction control conditions) or approximately 5 days (range = 3-7) after enrollment (care as usual condition)
  19-question assessment of anxiety specifically related to events surrounding a cesarean delivery. Score is 1-5 for each question. Minimum score 19. Maximum score 95.
Wijma Delivery Expectancy/Experience Questionnaire | Approximately 3 days (range=1-5) after intervention (CARE and interaction control conditions) or approximately 5 days (range = 3-7) after enrollment (care as usual condition)
  33-item measure of fear of childbirth expectancy. Higher scores are related to higher fear regarding childbirth. Minimum score 0. Maximum score 165.
Intervention and Interaction Control Acceptability | 3 weeks post-delivery
  Satisfaction with intervention session: Minimum score 1. Maximum score 5.
Cesarean Section Anxiety Sensitivity (C-SAS) | 3 weeks post-delivery
  19-question assessment of anxiety specifically related to events surrounding a cesarean delivery. Score is 1-5 for each question. Minimum score 19. Maximum score 95.
HCAHPS | 3 weeks post-delivery
  A 29-question standardized patient satisfaction survey is used across U.S. hospitals to measure patients' perspectives on their hospital experience. Minimum score 0. Maximum score 100, and higher scores express a more positive experience.
State-Trait Anxiety Inventory | 12 weeks post-delivery
  20-item scale to assess state anxiety symptom intensity. Higher scores indicate more intense anxiety symptoms. Minimum score 20. Maximum score 80.
Columbia Suicide Severity Rating Scale | 12 weeks post-delivery
  6-item scale to assess presence of suicidal ideation, plan and intent. With any yes answer indicating some form of suicidality.
Posttraumatic Stress Disorder Checklist-5 | 12 weeks post-delivery
  20-item scale to assess trauma symptoms associated with acute stress disorder and posttraumatic stress disorder. Higher scores indicate more trauma symptoms regarding childbirth. Minimum score 0. Maximum score 80.
Edinburgh postpartum depression scale | 12 weeks post-delivery
  10-item scale to assess the presence of depression symptoms in the perinatal period. Higher scores indicate higher incidence of depressive symptoms. Minimum score 0. Maximum score 30.
Wijma Delivery Expectancy/Experience Questionnaire | 12 weeks post-delivery
  33-item measure of fear of childbirth expectancy. Higher scores are related to higher fear regarding childbirth. Minimum score 0. Maximum score 165.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available to the scientific community on the date that the grant award period ends. Sharing of materials will be facilitated as part of the normal conduct of collaborative research. All terms will comply with published NIH guidelines for the dissemination of research resources. All resource tools generated in conjunction with this project will be distributed freely and shared with the scientific community via peer-reviewed publications and poster/oral presentations at national/international meetings. The investigators will also openly share unpublished results with the scientific community as opportunity presents and/or the data is requested.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be made available to the scientific community on the date that the grant award period ends. Sharing of materials will be facilitated as part of the normal conduct of collaborative research. All terms will comply with published NIH guidelines for the dissemination of research resources. All resource tools generated in conjunction with this project will be distributed freely and shared with the scientific community via peer-reviewed publications and poster/oral presentations at national/international meetings. The investigators will also openly share unpublished results with the scientific community as opportunities present and/or the data is requested.
Access Criteria: For all shared data, any interested reseacher can have access to this data through a data use agreement from the university of colorado.
URL: https://redcap.ucdenver.edu/surveys/index.php?s=LNXN9C3JM9